CLINICAL TRIAL: NCT02284061
Title: Physical Activity Program in Children and Adolescents With Cancer : Assessment of Benefits on Physical, Psychological and Social Health.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2014-25; APHM (Other: RCAPHM14_0204)
Record Dates: First submitted 2014-10-23; First posted 2014-11-05 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

ARMS (2):
- experimental (Experimental): Immediate Program : the child follows the physical activity program for a period of 18 months, as soon as his medical condition permits.
  Interventions: Other: physical activities adapted to children
- Control (Other): Delayed Program: the child does not participate to the program during the first 6 months, and he joins the delayed program late after 6 months.
  Interventions: Other: physical activities adapted to children

INTERVENTIONS:
Other: physical activities adapted to children

SUMMARY:
Context: Sport and physical activity during and after cancer treatment can improve fitness and social inclusion in adults. In children, although early studies show interesting results, conclusive data are lacking. A preliminary evaluation conducted in a dozen children following a physical training program showed a significant improvement in endurance, muscle tone, overall self-esteem, sports skills and self-perceived strength. The investigators then want to evaluate the health of a group of children during treat cancer that physical activities adapted compared to children who did not practice.

Objective: Measuring the impact of physical activity program on health of children and adolescents with cancer with improved physical, psychological health, social reintegration and reduced time hospitalization.

Method and Design: The study plans to include 90 children from the pediatric hematology - oncology department of the La Timone CHU, aged 5-19 years with cancer, over a period of 18 months.

This is a randomized controlled open trial open with a stratified distribution. Children will be randomized between two arms - Arm A (Experimental - Immediate Program): the child follows the physical activity program for a period of 18 months, as soon as his medical condition permits. - Arm B (Control - Delayed Program): the child does not participate to the program during the first 6 months, and he joins the delayed program late after 6 months. Each child integrates the physical program for a period of one year.

Regardless of the randomization arm, the child performs the initial tests, the intermediate tests at 6 and 12 months and final tests at 18 months. Follow-up physical testing will be performed at 3 and 9 months.

The physical activity program includes a minimum of 30 days of activities per 6 months (4days/month and a long stay). The child practice between 2 to 4 hours of activity per day.

The investigators aim at demonstrating a difference of 50 meters on the total walked distance during the endurance test in the experimental group as compared to the control group after 6 months of program.

ELIGIBILITY:
Inclusion Criteria:

* Patient with malignant disease
* Supported in service pediatric hematology-oncology child Timone hospital in Marseille.
* Age ≥ 5 years and ≤ 19 years
* No medical-cons to the practice of physical activity

Exclusion Criteria:

* Life expectancy less than 18 months.
* Inability to comply with follow-up study for geographical, social or psychological.
* Length of stay less than 18 months, for children living outside mainland
* Not understanding of the French language
* Prior Participation in physical activity program

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
change of 50 meters on the total walked distance during the endurance test in the experimental group as compared to the control group after 6 months of program. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — APHM
Locations (1):
- Assistance publique hopitaux de marseille, Marseille, France